CLINICAL TRIAL: NCT02747888
Title: Hereditary Risk Factors for Thyroid Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Junne Kamihara, MD, MD, PhD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15-159
Record Dates: First submitted 2016-03-31; First posted 2016-04-22 (Estimated); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Cancer
Keywords: Thyroid
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower Suspected Familial Predisposition (No Intervention): Lower Suspected Familial Predisposition
  Screening and Enrollment:
  Consent, Family HX, Medical HX, Blood/Saliva which will categorize by suspected hereditary predisposition: Based on family and medical history.
  - Sample stored in Biorepository
- Higher Suspected Familial Predisposition (Experimental): Higher Suspected Familial Predisposition
  Screening and Enrollment:
  Consent, Family HX, Medical HX, Blood/Saliva which will categorize by suspected hereditary predisposition: Based on family and medical history.
  - Specimen Testing and Analysis
  •Referral to Genetic Counselor, if indicated
  Interventions: Genetic: •Referral to Genetic Counselor, if indicated

INTERVENTIONS:
Genetic: •Referral to Genetic Counselor, if indicated
  Arms: Higher Suspected Familial Predisposition

SUMMARY:
Thyroid cancers can occur sporadically, but can also be found as tumors that cluster in families with other cancers or genetic syndromes. Researchers are studying thyroid cancer in children and families, with a particular interest in understanding genes and other factors that may put individuals at risk for developing thyroid cancer and thyroid nodules.

* In this study, family and medical history information is collected alongside a blood or saliva sample for genetic studies.
* Individuals with a past or present childhood thyroid cancer/nodule or a thyroid cancer suspected to be inherited in their family are invited to participate.

DETAILED DESCRIPTION:
The purpose of this research study is to learn more about risk factors for inherited thyroid cancer.

The investigators would like to use the participant DNA to look for alterations in genes. The investigator will perform DNA sequencing and other genetic studies to identify errors in the genes that may contribute to the formation of thyroid nodules and cancer.

ELIGIBILITY:
Inclusion Criteria:

* Individual pediatric patient with current or previous known or suspected thyroid cancer or nodule(s).
* Individual adult patient with current or previous known or suspected thyroid cancer or nodule(s) if they come from a family with a high suspicion of hereditary cancer (as below).
* Individuals from families with a high suspicion of hereditary thyroid cancer:

  * Families with a current or previous diagnosis of a thyroid cancer/nodule occurring in childhood (<18 years old).
  * Families with a high suspicion of hereditary thyroid cancer/nodules other than above to include:

    * Families with thyroid cancer in multiple individuals
    * Families with thyroid cancer and a known genetic syndrome
    * Families with thyroid cancer and a suspected genetic syndrome (e.g. multiple childhood cancers in the family, multiple primary cancers, multiple endocrinopathies, etc.)

Exclusion Criteria:

* Individuals who are unable to give informed consent.
* Individuals who are unable to complete study materials.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have childhood or suspected familial thyroid nodules/cancer | 2 years
Number of germline mutations identified associated with thyroid cancer predisposition | 2 years
Prevalence of suspected familial thyroid cancer among those with childhood thyroid nodules/cancer | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Junne Kamihara, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No